CLINICAL TRIAL: NCT00762840
Title: Clinical Study to Evaluate the Safety and Efficacy of the Apexum Ablator in Subjects With Periapical Lesions Associated With Root Canal Infection
Brief Title: Safety and Efficacy of the Apexum Ablator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Apexum Ltd. (Industry)
Collaborators: Monitoring: Quail CRO, Romania (Unknown); Medistat Ltd., Israel (Industry)
Responsible Party: Idan Tobis, General manager, Apexum Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Apexum Trial
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Periapical Periodontitis
Keywords: Periapical lesions; Apical Periodontitis; endodontic procedure; root canal treatment
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apexum (Experimental): the tooth is treated by a standard root canal treatment, supplemented by Apexum Ablator protocol, in which the periapical lesion tissue is minced and removed through the root canal, in a minimally invasive fashion.
  Interventions: Device: the Apexum Protocol; Procedure: Conventional endodontic procedure
- Control (Active Comparator): the tooth is subject to conventional endodontic procedure alone, (standard root canal treatment)
  Interventions: Procedure: Conventional endodontic procedure

INTERVENTIONS:
Device: the Apexum Protocol — using the apexum kit for minimally invasive removal of periapical lesion tissue.
  Arms: Apexum
Procedure: Conventional endodontic procedure — Standard root canal treatment

SUMMARY:
The study is designed to test the hypothesis that there is a difference in healing kinetics and healing rate between teeth treated by conventional endodontic procedure alone and those in which such procedure was supplemented with the Apexum Ablator protocol

DETAILED DESCRIPTION:
Periapical lesions consist of inflammatory tissue replacing the bone surrounding the root-tip (apex) and are caused by bacteria present in an infected root canal (Metzger 2000). Endodontic (root canal) treatment is performed to eliminate these bacteria from the root canal and prevent its recontamination. The periapical lesion is expected to heal in response to this procedure, with new bone replacing the soft tissue of the lesion. The healing of the lesion may last 6-48 months, depending on its size and individual healing rate (Wang et al 2004).

Not all lesions heal accordingly. Those which fail to heal are subjected to either non-surgical re-treatment or to a surgical procedure called "apicoectomy" (Kim & Kratchman 2006). The surgical procedure consists of cutting the gums, accessing the periapical tissue through a hole drilled in the cortical bone, followed by curetting the soft tissue out of its bony crypt. After such surgical procedure, bone healing is much quicker (Kvist & Reit 1999) and even relatively large lesions may heal within 3-6 months. Nevertheless, pain and swelling usually inflict great discomfort causing patients to lose up to 6 working days (Kvist & Reit 2000).

It is common practice to delay the final dental restoration (crown or bridge) for as long as the periapical lesion has not healed. Even though a surgical intervention could significantly reduce the waiting time, it is not commonly applied due to following: (a) Pain, discomfort and loss of working days, (b) High cost (c) Inaccessibility of many root tips, due to anatomical reasons.

Apexum has developed a family of miniature, minimally invasive surgical tools, facilitating highly innovative methods for the treatment of periapical lesions associated with root canal infection. The Apexum Ablator device allows access to the periapical tissues through the root-canal following the commonly accepted root-canal procedures. The inserted tool grinds the periapical lesion, followed by washing out and aspiration of the ground material.

In the present study, the safety and efficacy of the Apexum Ablator will be assessed in patients with periapical lesions associated with root canal infection by using this clinical investigational plan.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years old
2. Subject has periapical lesion(s) associated with root canal infection in one or more roots that have a single root canal per root. These may include upper and lower single rooted incisors, canines or premolars, as well as roots of multi-rooted teeth, providing that they have a single root canal per root. These may include distal roots of lower molars, palatal and disto-buccal roots of upper molars
3. Lesion mean diameter: 3-6 mm, PAI score 4 or 5
4. Roots with mature fully formed apices

Exclusion Criteria:

1. Previous root canal filling
2. Roots with abnormal root canal morphology
3. Roots with more than one root canal per root, as either evident from the pre-operative radiographs or as discovered during initiation of the root canal treatment
4. A tooth that remained symptomatic after the first and when needed a second session of the root canal treatment (remained with an excessive sensitivity to percussion, persistent sinus tract, persistent exudate in the root canal etc.)
5. Un-restorable teeth
6. Significant periodontal pockets
7. Lack of cortical bone around the lesion, as judged clinically
8. Active acute infection - cellulites, abcess
9. Proximity of anatomical structures to the periapical lesion to the extent that Apexum Ablator enucleation procedure may damage or otherwise jeopardize these structures. Such anatomical structures may include the maxillary sinus, the nasal cavity, the inferior alveolar nerve and its canal, the mental nerve or any other structure that may be jeopardized by the procedure
10. Subject with:

    * Uncontrolled systemic hypertension
    * Severe uncontrolled Diabetes Mellitus
    * Current steroid therapy in excess of prednisone 5 mg/day
    * Chronic inflammatory oral disease
    * HIV positive patients
    * Chronic renal failure
    * Hematological disease (malignancy, severe anemia, bleeding tendency etc.)
    * Osteoporosis, receiving biphosphonates
    * Post head and neck irradiation treatment
    * In need of endocarditis antibiotic prophylactic treatment [sub acute bacterial endocarditis (SBE]
11. Other severe or life-threatening systemic disease (ASA P3 and above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-10; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Healing at 6-month follow-up, defined dichotomously by whether lesion is in the process of Healing or not, indicated by whether PAI score at 6 months is at 3 or below | 6 months

SECONDARY OUTCOMES:
Healing at 12-month follow-up. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dragos Slavescu, DMD, Principal Investigator — Titu Maiorescu University; Dan Dragomirescu, DMD, Principal Investigator — Cabinet Stomatologic Dr Dan Dragomirescu
Locations (2):
- Romania (2):
  - Titu Maiorescu University, Bucharest
  - Cabinet Stomatologic Dr Dan Dragomirescu, Timișoara